CLINICAL TRIAL: NCT07115446
Title: A Phase Ib Study to Explore the Safety, Tolerability, and Pharmacokinetics of HS-20093 Combination With HRS-5041 in Patients With Advanced Prostate Cancer
Brief Title: Phase Ib Study of HS-20093+HRS-5041 in Patients With Advanced Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-20093-107
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Advanced Prostate Cancer
Keywords: Advanced prostate cancer; B7H3; HS-20093

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HS-20093+HRS-5041 (Experimental): Participants will receive HS-20093 at RP2D and HRS-5041 at Dose1 or Dose2.
  Interventions: Drug: HS-20093; Drug: HRS-5041

INTERVENTIONS:
Drug: HS-20093 — Intravenous (IV) administration of HS-20093 Q3W; Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.
Drug: HRS-5041 — HRS-5041 was given oral administration, QD, at a 21-day cycle.

SUMMARY:
HS-20093 is a fully humanized IgG1 antibody-drug conjugate (ADC) which specifically binds to B7-H3, a target wildly expressed on solid tumor cells. HRS-5041 is a Proteolysis Targeting Chimeras (PROTAC) targeting androgen receptors.

This is a phase Ib, open-label, multi-center study to evaluate the safety, tolerability, and pharmacokinetics (PK) of HS-20093 combination with HRS-5041 in patients with advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men greater than or equal to 18 years.
* Voluntarily to participate, Signed and dated Informed Consent Form.
* Patients with metastatic castration-resistant prostate cancer (mCRPC) who progressed after at least one type of novel hormonal therapy (standard treatment).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0~1.
* Estimated life expectancy ≥ 12 weeks.
* Men should use adequate contraceptive measures throughout the study, up to 3 months after the last dose of HRS-5041 or 4.5 months after the last dose of HS-20093 (whichever is later).

Exclusion Criteria:

* Treatment with any of the following:

  a. Previous or current treatment with B7-H3 targeted therapy. b. Previous treatment with AR PROTAC. c. Any cytotoxic chemotherapy, investigational agents and anticancer drugs within 21 days prior to the first scheduled dose of HS-20093+HRS-5041. d. brain metastases.
* Any unresolved toxicities from prior therapy greater than Grade 2 according to Common Terminology Criteria for Adverse Events (CTCAE) 5.0.
* History of other primary malignancies.
* Inadequate bone marrow reserve or organ dysfunction.
* Severe, uncontrolled or active cardiovascular diseases.
* Severe or uncontrolled diabetes.
* The presence of active infectious diseases.
* Any known or suspected interstitial lung disease.
* History of serious neuropathy or mental disorders.
* History of severe hypersensitivity reaction, severe infusion reaction.
* Hypersensitivity to any ingredient of HS-20093.
* Unlikely to comply with study procedures, restrictions, and requirements in the opinion of the investigator.
* Any disease or condition that, in the opinion of the investigator, would compromise subject safety or interfere with study assessments.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) or Maximum Administrated dose (MAD) | 21 days from administration of the first dose (C1D1) in the dose escalation phase， assessed up to 24 months
  Number of participants with dose limiting toxicity

SECONDARY OUTCOMES:
To evaluate the incidence and severity of adverse events (AEs) | From the first dose(C1D1) up to 30 days after the last dose of HRS-5041 or 90 days after the last dose of HS-20093 (whichever is later)
  AE assessed by investigator exclusively related to subject's underlying disease or medical condition [graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0]. Any untoward medical occurrence in a participant, whether or not considered related to the medicinal product. Incidence and severity of AEs are assessed according to vital signs, laboratory variables, physical examination, electrocardiogram, etc.
To evaluate the maximum plasma concentration (Cmax) | up to approximately 24 months
  Cmax will be obtained following administration of the first dose of HS-20093 during the first cycle
To evaluate the Time to reach maximum plasma concentration (Tmax) | up to approximately 24 months
  Tmax will be obtained following administration of the first dose of HS-20093 during the first cycle
To evaluate the Area under plasma concentration versus time curve from zero to last sampling time (AUC) | up to approximately 24 months
  Area under the plasma concentration versus time curve from time zero to the last sampling time when the concentration was no less than the lower limit of quantification (LLQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule
To evaluate the immunogenicity of HS-20093 | up to approximately 24 months
  Proportion of patients who are positive for anti-HS-20093 antibodies
To evaluate the ORR determined by investigators | up to approximately 24 months
  Objective response rate (ORR) determined by IRC according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and Prostate Cancer Working Group 3 (PCWG3)
To evaluate the Disease control rate (DCR) determined by investigators according to RECIST 1.1 and PCWG3 | up to approximately 24 months
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). DCR was evaluated by the number of participants with best overall response of CR, PR and stable disease (SD) [Confirmed CR/PR assessment require at least one repeat (≥4 weeks); SD shall be assessed at least 5 weeks after the first dose]
To evaluate the Duration of response (DoR) determined by investigators according to RECIST 1.1 and PCWG3 | up to approximately 24 months
  DoR is defined as the period from the first occurrence of CR or PR to progressive disease (PD) or death from any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) would be used [Confirmed CR/PR assessment require at least one repeat (≥4 weeks)]
To evaluate the Prostate-specific Cancer Antigen (PSA) response rate（PSA30,PSA50,PSA90） | up to approximately 24 months
  PSA response is defined as a ≥ 30%，≥ 50% ，≥ 90% decline in PSA from baseline with PSA confirmation ≥ 3 weeks after the first documented reduction
To evaluate the Time to PSA progression | up to approximately 24 months
  In participants with a decrease in PSA from baseline: ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the nadir value, which is confirmed by a consecutive second value obtained ≥ 3 weeks later. In participants with no decrease in PSA from baseline: ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the baseline value after 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China